CLINICAL TRIAL: NCT02729584
Title: Gene Polymorphism of Taste Receptors and Circulating Endocannabinoids in Normal Weight and Obese Subjects
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Ospedaliera Brotzu (Other)
Responsible Party: Principal Investigator, Sebastiano Banni, Professor, University of Cagliari
Other Study IDs: Cagliari
Record Dates: First submitted 2016-03-23; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Nutritional Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight
- Obese

SUMMARY:
The study aims at evaluating in normal weight and obese subjects those factors such as taste sensitivity and circulating endocannabinoids in influencing dietary choice and thereby lipid and energy metabolism in order to design personalized nutritional strategies.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI), range for normal weight subjects 17.5-24.95, for obese subjects 29.6-52.20
* No intake of nutritional supplements for at least six months before the trial

Exclusion Criteria:

* major diseases (diabetes, kidney disease, etc.),
* pregnancy or lactation;
* food allergies;
* the use of medications that interfere with taste or smell (e.g., steroids, antihistamines, certain antidepressants).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: White Caucasians
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Endocannabinoid plasma levels | 1 year

IPD SHARING:
Plan to Share IPD: No